CLINICAL TRIAL: NCT07387302
Title: A Phase II Clinical Study Evaluating SLN12140 in Complement Inhibitor-Naïve Adult Subjects With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: SLN12140 in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) in China
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Linno Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIN2102-CN201
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SLN 12140 will be administered subcutaneously . (Experimental): 5 participants will receive SLN12140 100mg QW for 4 weeks, then 300mg QW for 8 weeks, then 200mg QW for 52 weeks.
  5 participants will receive SLN12140 200mg QW for 4 weeks, then 600mg Q4W for 60 weeks
  Interventions: Drug: SLN12140

INTERVENTIONS:
Drug: SLN12140 — 5 participants will receive SLN12140 100mg QW for 4 weeks, then 300mg QW for 8 weeks, then 200mg QW for 52 weeks. 5 participants will receive SLN12140 200mg QW for 4 weeks, then 600mg Q4W for 60 weeks

SUMMARY:
The goal of this clinical trial is to learn if drug SLN12140 works to treat Complement Inhibitor-Naïve Subjects with Paroxysmal Nocturnal Hemoglobinuria in adults. It will also learn about the safety, pharmacokinetic characteristics, and dosing of drug SLN12140.

The study is divided into four phases: screening period, core treatment period, extended dosing period, and follow-up period, and includes two cohorts (Cohorts 1-2), with each cohort enrolling at least 5 treatment-naïve adult PNH subjects for complement inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult complement inhibitor naïve PNH patients (age>=18), which is confirmed by flow cytometry evaluation
* Must be vaccinated against meningococcal vaccine and pneumococcal vaccine

Exclusion Criteria:

* Significant bone marrow failure
* Meningitidis infection or unresolved meningococcal disease
* Other significant systemic diseases that might have impact on efficacy and safety assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
During the 12-week treatment period, the proportion of participants whose Lactate Dehydrogenase (LDH) decreased by 60% or more from baseline or whose LDH was below the upper limit | 12weeks after baseline
  To assess efficacy of SLN12140 in participants with PNH

SECONDARY OUTCOMES:
Percentage change of LDH from baseline | Baseline through Week 64
  To assess the efficacy of SLN12140 in participants with PNH
Proportion of participants achieving hemolysis control (LDH ≤ 1.5×ULN) | Baseline through Week 64
  To assess the efficacy of SLN12140 in participants with PNH
Change in hemoglobin (Hb) levels from baseline | Baseline through week 64
  To assess the efficacy of SLN12140 in participants with PNH
The proportion of participants whose hemoglobin (Hb) increased by ≥2 g/dL from baseline and who avoided blood transfusion | Baseline through Week 64
  To assess the efficacy of SLN12140 in participants with PNH
Proportion of participants who avoided blood transfusion | Baseline through Week 64
  To assess the efficacy of SLN12140 in participants with PNH
Incidence(%) of Breakthrough Hemolysis (BTH) | Baseline through Week 64
  To assess the efficacy of SLN12140 in participants with PNH
Changes from baseline in intravascular and extravascular hemolysis indicators (including but not limited to reticulocytes, bilirubin, red blood cell count, platelet count, ferritin, etc.) | baseline through week 64
  To assess the efficacy of SLN12140 in participants with PNH
Changes in thrombus formation risk markers from baseline (including but not limited to fibrinogen, prothrombin time, activated partial thromboplastin time, thrombin time, fibrin D-dimer, etc.); | Baseline through week 64
  To assess the efficacy of SLN12140 in participants with PNH
Change in functional assessment of Functional Assessment of Chronic Illness Therapy (FACIT) | Baseline through Week 64
  To assess the efficacy of SLN12140 in participants with PNH. FACIT is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function to assess the Impact of SLN12140 on Treatment-Related Outcomes. The minimum value is 0 and maximum value is 52, and higher scores mean a worse outcome.
Number(%) of participants with Adverse Events (AEs) , Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline through Week 64
  To assess the safety and tolerability of SLN12140 in participants with PNH
Pharmacokinetics (PK)parameters of SLN12140: Area Under The Plasma Concentration-time Curve | Baseline through week 64 (predose and postdose)
  To characterize the pharmacokinetics of SLN12140 in participants with PNH
Immunegenicity in Paraxysmal Nocturnal Hemoglobinuria | Baseline through Week 64
  Determine anti-drug antibody titers
PK: Maximum Plasma Concentration (Cmax) | Baseline through week 64( predose and postdose)
  To characterize the pharmacokinetics of SLN12140 in participants with PNH
PK: Time To Maximum Concentration (Tmax) | Baseline through week 64( predose and postdose)
  To characterize the pharmacokinetics of SLN12140 in participants with PNH
Complement Alternative Pathway (AP) Functional Activity | Baseline through week 64( predose and post dose)
  Serum AP functional activity was measured by the Wieslab functional immunoassay method.
Complement FP | Baseline through week 64(predose and postdose)
  Plasma FP was measured by enzyme-linked immunosorbent assay (ELISA).

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided yet at this moment if we will share IPD with other researchers, or when will IPD will be shared, or with whom will IPD be shared, or by what mechanism will IPD be shared.